CLINICAL TRIAL: NCT00428896
Title: A Pilot Feasibility Study to Evaluate the Efficacy of ZD1839 (IRESSA) in Eliminating Chemo- and Hormone- Resistant Cytokeratin-Positive Tumour Cells Circulating in the Blood of Women With Breast Cancer
Brief Title: A Feasibility Study With Iressa in Resistant Cytokeratin-Positive Tumor Cells Circulating in the Blood of Women With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of Crete (Other)
Responsible Party: V.Georgoulias, University Hospital of Crete
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MICRO
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2008-07-21 (Estimated); Status verified 2008-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; iressa circulating tumor cells
MeSH Terms: conditions — Breast Neoplasms | interventions — Gefitinib

ARMS (1):
- 1 (Experimental): ZD1839
  Interventions: Drug: ZD1839

INTERVENTIONS:
Drug: ZD1839 — ZD1839 will be given at the dose of 250mg/day for a minimum of 3 months
  Other Names: Iressa

SUMMARY:
Based on preclinical data, ZD1839 is considered a novel and promising therapeutic approach with potential application in the treatment of human breast cancer. Therefore it could be very important and clinically relevant to know if ZD1839 is capable of eliminating occult tumour cells circulating in the blood of breast cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Histologically or cytologically confirmed breast cancer
* Metastatic breast cancer (stage IIIB and IV)
* Patients should have received at least one course of standard systemic chemotherapy for their metastatic disease. There should be at least one month between end of chemotherapy treatment and trial entry.
* ER+ve patients should have received adjuvant hormonal treatment
* Detection of CK-19 mRNA positive cells in the blood by real time PCR despite the previous administration of chemotherapy and if appropriate hormonal therapy
* Aged 18 years and over
* Paraffin-embedded tissue available for tumour histology (EGFR testing, ER, PgR, Her-2-neu testing)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2
* Patients willing to undergo regular detection of circulating occult tumour cells in the blood by immunocytochemistry and/or RT-PCR
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Any concurrent systemic treatment for breast cancer (including chemotherapy, radiotherapy, hormonotherapy, monoclonal antibodies)
* Known severe hypersensitivity to ZD1839 or any of the excipients of this product
* Any evidence of clinically active interstitial lung disease (patients with chronic, stable, radiographic changes who are asymptomatic need not be excluded)
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Any unresolved chronic toxicity greater than common toxicity criteria (CTC) grade 2 from previous anticancer therapy (except alopecia)
* Serum bilirubin greater than 1.5 times the upper limit of reference range (ULRR)
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* Alanine amino transferase (ALT) or aspartate amino transferase (AST) greater than 3 times the ULRR.
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study
* Pregnancy or breast feeding (women of child-bearing potential). Women of childbearing potential must practice acceptable methods of birth control to prevent pregnancy
* Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St John's Wort
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of ZD1839 by quantitative analysis of CK-19 mRNA CTCs | Detection of CK-19 mRNA CTCs during and after the completion of ZD1839 treatment

SECONDARY OUTCOMES:
To assess duration of response by means of CK-19 mRNA detection | 6 months
To assess Progression Free Survival by means of CK-19 mRNA detection | 1 year
To assess the safety of ZD1839 administration in this patient population | Toxicity assessment every month

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (1):
- University Hospital of Crete, Heraklion, Crete, Greece

REFERENCES:
- [Derived] Kalykaki A, Agelaki S, Kallergi G, Xyrafas A, Mavroudis D, Georgoulias V. Elimination of EGFR-expressing circulating tumor cells in patients with metastatic breast cancer treated with gefitinib. Cancer Chemother Pharmacol. 2014 Apr;73(4):685-93. doi: 10.1007/s00280-014-2387-y. Epub 2014 Feb 4. PMID 24493157